CLINICAL TRIAL: NCT03490331
Title: Prospective, Open-label, Uncontrolled Clinical Trial to Assess the Safety and Efficacy of Autologous Cultured Epidermal Grafts Containing Epidermal Stem Cells Genetically Modified With a Gamma-retroviral (rv) Vector Carrying COL17A1 cDNA for Restoration of Epidermis in Patients With Junctional Epidermolysis Bullosa
Brief Title: Clinical Trial to Assess Safety and Efficacy of Autologous Cultured Epidermal Grafts Containing Epidermal Stem Cells Genetically Modified in Patients With JEB (HOLOGENE17)
Acronym: HOLOGENE17
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No patient ongoing (none completed the study). Changes to the viral vector ongoing.
Sponsor: Holostem s.r.l. (Industry)
Collaborators: Paracelsus Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTA-HG17-01
Record Dates: First submitted 2018-03-18; First posted 2018-04-06 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Junctional Epidermolysis Bullosa
Keywords: JEB; Stem cells; Gene Therapy
MeSH Terms: conditions — Epidermolysis Bullosa, Junctional | interventions — cyclic adenosine-5'-trimetaphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genetically corrected cultured epidermal autograft (Experimental): The surgery will be carried out in 2 stages, the first aims at taking biopsy to isolate epidermal cells including stem cells. The biopsy will be processed in a laboratory of a regenerative medicine manufacturing site where they will be corrected, expanded and prepared as final sheets to be implanted.
  In the second surgery, genetically corrected cultured epidermal autograft (Hologene17) will be implanted into the selected area. The specialist surgeon will either use a local or general anaesthetic for the implant operation. The treated area will be immobilized for some days after this operation. Antibiotics and anti-inflammatory drugs will be administered (if necessary) to prevent infections and to minimise swelling.
  Interventions: Other: Transplantation surgery of genetically corrected cultured epidermal autograft (ATMP)

INTERVENTIONS:
Other: Transplantation surgery of genetically corrected cultured epidermal autograft (ATMP) — Surgergical procedure for transplantation under anaesthesia of genetically corrected cultured epidermal autograft (Hologene17) on blistering skin areas of JEB patients. By taking some autologous epidermal cells, a new layer of transgenic tissue is grown in the laboratory. This layer of tissue - containing genetically modified stem cells - is then implanted by a surgeon into the damaged area. The implantation can be done in one or more areas and repeated in case of failure of the first surgery.
  Other Names: Transplantation of Hologene17 study product (ATMP)

SUMMARY:
Prospective open-label, uncontrolled clinical study to assess the safety and efficacy of autologous cultured epidermal grafts containing epidermal stem cells genetically modified with the aid of a gamma-retroviral vector carrying COL17A1 complementary DNA (cDNA) for restoration of the epidermis in patients with junctional epidermolysis bullosa. The purpose of this study is to demonstrate the safety and efficacy after one or more treatments with genetically corrected cultured epidermal autograft (Hologene 17) in patients suffering of junctional epidermolysis bullosa (JEB) with COL17A1 mutation.

DETAILED DESCRIPTION:
This is a prospective, open label, uncontrolled clinical trial, phase I/II. Patients will be screened according to the Study Inclusion and Exclusion criteria and will be candidate for the treatment if all inclusion and none of the exclusion criteria are met.

After confirmation of eligibility, patients will undergo biopsy for the collection of the autologous epidermal cells to be used to produce the tissue for the treatment. In case all criteria are met, the transplantation of the new cultured transgenic epidermis will be planned according to the procedures and the need of the patient.

The study treatment consists of a surgical intervention for new restored stem cells implantation.

The surgery will be carried out in 2 stages, the first aims at taking biopsy to isolate epidermal cells including stem cells. The biopsy will be processed in a laboratory of a regenerative medicine manufacturing site where they will be corrected, expanded and prepared as final sheets to be implanted. Therefore, the patient can have his second intervention. In this second surgery, genetically corrected cultured epidermal autograft (Hologene 17) will be implanted into the selected area. The specialist surgeon will either use a local or general anaesthetic for the transplant operation. The treated area will be immobilized for some days after this operation. Antibiotics and anti-inflammatory drugs will be administered (if necessary) to prevent infections and to minimise swelling.

Three months after the transplantation, primary endpoint will be evaluated by the Investigator. The study completion will be reached when 1 year (secondary endpoint) of follow-up after the last transplant in the last patient will be accomplished.

The end of the trial is defined as the last visit of the last patient after the last treatment if any.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent prior to any study-related procedures;
2. Male and female patients between 6 years old to 54 years old;
3. JEB molecular characterization by mutation analysis;
4. NC16A antibody immunofluorescence or positive staining in Western Blot analysis with polyclonal antibody produced against a synthetic peptide corresponding to amino acids 131-145 of human COL17A1;
5. Presence of chronic (persistent or recurrent for more than 3 months) large wounds (>10 cm2) and/or persistent or recurrent erosions;
6. A cooperative attitude to follow up the study procedures (Caregivers in case of minors).

Exclusion Criteria:

1. Known or suspected intolerances against anaesthesia;
2. Bad general condition (ECOG index >1);
3. Unresectable metastasizing Squamous Cell Carcinomas (SCCs);
4. Antibodies to type XVII collagen associated antigens demonstrated on indirect immunofluorescence;
5. Clinical and/or laboratory signs of acute systemic infections at the time of screening. Patient can be re-screened after appropriate treatment;
6. Severe systemic diseases (i.e. uncompensated diabetes mellitus);
7. Female subjects: pregnant or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential) UNLESS they are willing to use one or more reliable methods of contraception with a Pearl index ≤1. Reliable contraception should be maintained throughout the study.
8. Allergy, sensitivity or intolerance to drugs, excipients or other material (as per Investigator's brochure):

   * Transport medium (Dulbecco's Modified Eagles Medium supplemented with L-glutamine)
   * Fibrin support
   * Povidone iodine
9. Contraindications to the local or systemic antibiotics and/ or corticosteroids foreseen by the protocol;
10. Contraindications to undergo extensive surgical procedures;
11. Clinically significant or unstable concurrent disease or other clinical contraindications to stem cell transplantation based upon investigator's judgment or other concomitant medical conditions affecting grafting procedure;
12. Patients (or parents in case of paediatric subject) unlikely to comply with the study protocol or unable to understand the nature and scope of the study or the possible benefits or unwanted effects of the study procedures and treatments;
13. Participation in another clinical trial where investigational drug was received less than 6 months prior to screening Visit.

Ages: 6 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Safety events (ADRs and SAEs) related to the study treatment (tolerability) | 3 months after treatment
  Number of patients experiencing treatment-related adverse events (TRAEs) - either to the epidermal graft and to the surgical procedures. Adverse events (serious and not serious) and adverse drug reactions (ADRs) will be collected and described
Safety events (ADRs and SAEs) related to the study treatment (tolerability) | 12 months after treatment
  Percentage of patients experiencing treatment-related adverse events (TRAEs) - either to the epidermal graft and to the surgical procedures. Adverse events (serious and not serious) and adverse drug reactions (ADRs) will be collected and described

SECONDARY OUTCOMES:
Skin stability in the short term (Treatment efficacy) | 3 months after transplantation
  The skin stability will be evaluated by means of stripping test and visual inspection of the treated areas
Skin functionality in the short term (Treatment efficacy) | 3 months after transplantation
  The skin functionality will be evaluated by means of molecular testing on skin punch biopsies taken from the transplanted areas.
Skin stability in the long term (Treatment efficacy) | 12 months after transplantation
  The skin stability will be evaluated by means of stripping test and visual inspection of the treated areas
Skin functionality in the long term (Treatment efficacy) | 12 months after transplantation
  The skin functionality will be evaluated by means of molecular testing on skin punch biopsies taken from the transplanted areas.

CONTACTS AND LOCATIONS:
Overall Officials: Michele De Luca, MD/Professor, Study Director — Holostem s.r.l.; Johann W. Bauer, MD, Principal Investigator — Paracelsus Medical University - EB House
Locations (1):
- EB House Austria, Department of Dermatology, Paracelsus Medical University, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Correction of junctional epidermolysis bullosa by transplantation of genetically modified epidermal stem cells. — https://www.ncbi.nlm.nih.gov/pubmed/17115047
- See also: Description Long-term stability and safety of transgenic cultured epidermal stem cells in gene therapy of junctional epidermolysis bullosa. — http://www.ncbi.nlm.nih.gov/pubmed/24511464
- See also: Regeneration of the entire human epidermis using transgenic stem cells — http://www.nature.com/articles/nature24487
- See also: Description Closure of a large chronic wound through transplantation of gene-corrected epidermal stem cells. — http://www.ncbi.nlm.nih.gov/pubmed/27840234